CLINICAL TRIAL: NCT02206282
Title: Prevalence of Asymptomatic Rupture in SILIMED Breast Implants
Status: Completed | Type: Observational
Sponsor: Silimed Industria de Implantes Ltda (Industry)
Responsible Party: Sponsor
Other Study IDs: IMR-LT-001
Record Dates: First submitted 2014-07-28; First posted 2014-08-01 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Breast Implant Rupture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
A prospective clinical research is to assess the prevalence of implant rupture and presence of extracapsular gel in an un-referred population of women who have been implanted with the Silimed gel-filled mammary implants with or without any local or systemic systemic symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Subject implanted with the original Silimed gel-filled implant.

Exclusion Criteria:

* MR imaging is not possible because of the following:
* Metal implant
* Battery activated stimulator
* Pregnancy
* Tattoos
* Body weight >300 pounds
* History of metal fragments in the eye
* Any other contraindication to MR exam.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 390 women (780 implants) from Rio de Janeiro and other Brazilian cities will be randomly selected to undergo MRI detection of asymptomatic rupture using a stratified sampling design, stratifying on implant age (time since implantation). Sixty-five (65) women will be selected from each of six implant age groups between 6-18 years.
Sampling Method: Probability Sample
Enrollment: 390 (Actual)
Dates: Start 2006-08; Primary Completion 2010-11 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Magnetic Resonance Image | 1 year
  390 Magnetic Resonance Images.

CONTACTS AND LOCATIONS:
Overall Officials: Wanda Elizabeth Massiere Correa, MD, Principal Investigator — Insituto Ivo Pitanguy